CLINICAL TRIAL: NCT00690573
Title: A Multicenter, Open-label Study of the Safety, Efficacy, and Pharmacokinetics of the Human Anti-TNF Monoclonal Antibody Adalimumab in Children With Polyarticular Juvenile Rheumatoid Arthritis
Brief Title: Safety, Efficacy, and Pharmacokinetics of Adalimumab in Japanese Children With Juvenile Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-240
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2011-04-01 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab administered subcutaneously every other week, with dosage determined by body weight at study entry (20 mg for children weighing less than 30 kg, 40 mg for children weighing 30 kg or more).
  Other Names: adalimumab, ABT-D2E7, Humira

SUMMARY:
To evaluate efficacy, safety and pharmacokinetics of adalimumab in Japanese children with Polyarticular Juvenile Rheumatoid Arthritis

DETAILED DESCRIPTION:
This was an open-label long-term study that was completed following study drug approval in Japan for the treatment of JRA. Data are presented through Week 144 and for the final visit.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of polyarticular juvenile rheumatoid arthritis (JRA) according to the criteria of the American College on Rheumatology (ACR)
* Disease activity inadequately controlled by nonsteroidal anti-inflammatory drugs (NSAIDs) or methotrexate (MTX)
* Presence at screening of at least 5 swollen joints (not due to deformity) and at least 3 joints with limitation of passive motion with pain by passive motion or/and pain by pressure (tenderness)
* Stable dosage of MTX for at least 12 weeks prior to the screening visit or discontinuation of MTX at least 14 days prior to baseline visit (Day 1)
* Discontinuation of disease-modifying antirheumatic drugs (DMARDs) other than MTX at least 28 days before screening visit

Exclusion Criteria

* History of inflammatory joint disease other than JRA
* Functional class IV JRA by ACR criteria
* Clinically significant cardiac disease or laboratory abnormalities
* Any subject who is considered by the investigator, for any reason, to be an unsuitable candidate for the study

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, PhD, Study Director — Abbott Japan Co.,Ltd
Locations (12):
- Japan (12):
  - Site Reference ID/Investigator# 47248, Aichi
  - Site Reference ID/Investigator# 47253, Fukuoka
  - Site Reference ID/Investigator# 47251, Hyōgo
  - Site Reference ID/Investigator# 47254, Kagoshima
  - Site Reference ID/Investigator# 47250, Kobe
  - Site Reference ID/Investigator# 47255, Okinawa
  - Site Reference ID/Investigator# 7153, Sendai
  - Site Reference ID/Investigator# 47249, Takatsuki
  - Site Reference ID/Investigator# 47243, Tokyo
  - Site Reference ID/Investigator# 47244, Tokyo
  - Site Reference ID/Investigator# 47245, Tokyo
  - Site Reference ID/Investigator# 47246, Yokohama

REFERENCES:
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- [Derived] Imagawa T, Takei S, Umebayashi H, Yamaguchi K, Itoh Y, Kawai T, Iwata N, Murata T, Okafuji I, Miyoshi M, Onoe Y, Kawano Y, Kinjo N, Mori M, Mozaffarian N, Kupper H, Santra S, Patel G, Kawai S, Yokota S. Efficacy, pharmacokinetics, and safety of adalimumab in pediatric patients with juvenile idiopathic arthritis in Japan. Clin Rheumatol. 2012 Dec;31(12):1713-21. doi: 10.1007/s10067-012-2082-5. Epub 2012 Oct 2. PMID 23053683

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Adalimumab dose was determined by baseline body weight (20 mg for subjects weighing < 30 kg, 40 mg for subjects weighing 30 kg or more) through Week 14. After Week 16, dose was based on body weight measured at Week 16 and every 12 weeks. Twenty subjects received concomitant methotrexate therapy during the study.
Period: Overall Study
Arm/Group | Adalimumab
Started | 25
Completed | 16
Not Completed | 9
Not completed — Lack of Efficacy | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.0 (3.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Region of Enrollment [Number; unit: participants]
  Japan | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Pediatric American College of Rheumatology 30% (PedACR30) Response at Week 16
Description: Response defined as at least 30% improvement in 3 or more of 6 juvenile rheumatoid arthritis (JRA) core set criteria, and at least 30% worsening in not more than 1 JRA criterion, compared with baseline. JRA core set criteria include physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with limitation of motion [LOM] and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein.
Time Frame: Week 16
Population: The analysis was conducted using the full analysis set (FAS) population, which was defined as all subjects who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
Participants | 23

2. Secondary Outcome: Number of Subjects Achieving PedACR50 and PedACR70 Responses at Week 16
Description: Response defined as at least 50/70% improvement in 3 or more of 6 juvenile rheumatoid arthritis (JRA) core set criteria, and at least 50/70% worsening in not more than 1 JRA criterion compared with baseline. JRA core set criteria include physician's global assessment of disease severity; parent's/patient's global assessment of overall well-being; number of active joints (joints with swelling or with limitation of motion [LOM] and with pain, tenderness or both); number of joints with LOM; physical function of the Disability Index of Childhood Health Assessment Questionnaire; C-reactive protein.
Time Frame: Week 16
Population: The analysis was conducted using the full analysis set (FAS) population, which was defined as all subjects who received at least one dose of study drug. Missing values were treated as non-responders.
Measure: Number; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
Participants
  Number of Subjects Achieving PedACR50 at Week 16 | 22
  Number of Subjects Achieving PedACR70 at Week 16 | 15

3. Secondary Outcome: Number of Subjects Achieving PedACR 30/50/70 Responses
Time Frame: Week 2, 4, 8, and 24, every 12 weeks from Week 24 to Week 60, and every 24 weeks from Week 72 to the final visit
Population: The analysis was conducted using the full analysis set (FAS) population (all subjects who received at least 1 dose of study drug) as observed. N=25 at Weeks 2, 4, and the Final Visit; N=24 at Weeks 8, 24, and 36; N=23 at Week 48; N=22 at Week 60; N=19 at Weeks 72 and 96; N=11 at Week 120; and N=5 at Week 144.
Measure: Number; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
Participants
  Number of subjects achieving PedACR30 at Week 2 | 15
  Number of subjects achieving PedACR30 at Week 4 | 16
  Number of subjects achieving PedACR30 at Week 8 | 19
  Number of subjects achieving PedACR30 at Week 24 | 21
  Number of subjects achieving PedACR30 at Week 36 | 22
  Number of subjects achieving PedACR30 at Week 48 | 21
  Number of subjects achieving PedACR30 at Week 60 | 20
  Number of subjects achieving PedACR30 at Week 72 | 19
  Number of subjects achieving PedACR30 at Week 96 | 18
  Number of subjects achieving PedACR30 at Week 120 | 11
  Number of subjects achieving PedACR30 at Week 144 | 5
  Number of subjects achieving PedACR30- Final Visit | 22
  Number of subjects achieving PedACR50 at Week 2 | 7
  Number of subjects achieving PedACR50 at Week 4 | 13
  Number of subjects achieving PedACR50 at Week 8 | 15
  Number of subjects achieving PedACR50 at Week 24 | 19
  Number of subjects achieving PedACR50 at Week 36 | 22
  Number of subjects achieving PedACR50 at Week 48 | 19
  Number of subjects achieving PedACR50 at Week 60 | 20
  Number of subjects achieving PedACR50 at Week 72 | 18
  Number of subjects achieving PedACR50 at Week 96 | 18
  Number of subjects achieving PedACR50 at Week 120 | 11
  Number of subjects achieving PedACR50 at Week 144 | 5
  Number of subjects achieving PedACR50- Final Visit | 20
  Number of subjects achieving PedACR70 at Week 2 | 1
  Number of subjects achieving PedACR70 at Week 4 | 7
  Number of subjects achieving PedACR70 at Week 8 | 8
  Number of subjects achieving PedACR70 at Week 24 | 15
  Number of subjects achieving PedACR70 at Week 36 | 19
  Number of subjects achieving PedACR70 at Week 48 | 17
  Number of subjects achieving PedACR70 at Week 60 | 16
  Number of subjects achieving PedACR70 at Week 72 | 15
  Number of subjects achieving PedACR70 at Week 96 | 14
  Number of subjects achieving PedACR70 at Week 120 | 11
  Number of subjects achieving PedACR70 at Week 144 | 5
  Number of subjects achieving PedACR70- Final Visit | 17

4. Secondary Outcome: Mean Serum Adalimumab Concentration
Description: Blood samples were drawn prior to drug administration. Adalimumab concentrations in serum were determined using a validated enzyme-linked immunosorbent assay (ELISA) method based on a double-antigen technique. Concentrations are reported as micrograms per milliliter (mcg/mL).
Time Frame: Week 2, 4, 8, 16, and 24, and every 12 weeks up to Week 60
Population: For the 20 mg dose, N = 8 at each timepoint. For the 40 mg dose, N = 17 at Weeks 2 and 4; N = 16 at Weeks 8, 16, and 24; N = 14 at Week 36; N = 15 at Week 48; and N = 14 at Week 60.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
mcg/mL
  20 mg dose at Week 2 | 5.24 (1.74)
  20 mg dose at Week 4 | 5.46 (5.18)
  20 mg dose at Week 8 | 6.15 (5.88)
  20 mg dose at Week 16 | 5.73 (5.26)
  20 mg dose at Week 24 | 5.79 (6.51)
  20 mg dose at Week 36 | 7.60 (7.58)
  20 mg dose at Week 48 | 7.97 (6.69)
  20 mg dose at Week 60 | 11.4 (9.87)
  40 mg dose at Week 2 | 5.03 (1.45)
  40 mg dose at Week 4 | 5.63 (2.71)
  40 mg dose at Week 8 | 8.66 (4.41)
  40 mg dose at Week 16 | 10.8 (6.15)
  40 mg dose at Week 24 | 11.9 (6.80)
  40 mg dose at Week 36 | 12.6 (6.44)
  40 mg dose at Week 48 | 13.0 (8.89)
  40 mg dose at Week 60 | 13.1 (6.73)

5. Secondary Outcome: Number of Subjects Positive for Anti-adalimumab Antibodies (AAA)
Description: Serum samples with adalimumab concentration below 2 mcg/mL were selected for AAA analyses. Samples were considered AAA positive if the measured AAA concentration was above 20 ng/mL. A subject was considered to be AAA positive if the subject had at least one AAA positive sample observed within 30 days following the subject's last adalimumab dose.
Time Frame: Week 24 and Week 60
Measure: Number; unit: Participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 25
Participants
  Number of subjects with AAA by Week 24 | 4
  Number of subjects with AAA by Week 60 | 6

ADVERSE EVENTS:
Time Frame: All adverse events reported from the time of first study drug administration until 70 days following discontinuation of study drug administration were collected.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=25)
pyrexia (General disorders) | 2
hepatitis B (Infections and infestations) | 1
herpes zoster (Infections and infestations) | 1
pharyngitis (Infections and infestations) | 1
pneumonia (Infections and infestations) | 1
dehydration (Metabolism and nutrition disorders) | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1
juvenile arthritis (Musculoskeletal and connective tissue disorders) | 1
amnesia (Nervous system disorders) | 1
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=25)
iron deficiency anaemia (Blood and lymphatic system disorders) | 5
conjunctivitis (Eye disorders) | 2
conjunctivitis allergic (Eye disorders) | 3
keratoconjunctivitis sicca (Eye disorders) | 2
abdominal pain (Gastrointestinal disorders) | 3
abdominal pain upper (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 3
dental caries (Gastrointestinal disorders) | 3
diarrhoea (Gastrointestinal disorders) | 3
nausea (Gastrointestinal disorders) | 3
stomatitis (Gastrointestinal disorders) | 2
vomiting (Gastrointestinal disorders) | 2
injection site erythema (General disorders) | 4
injection site reaction (General disorders) | 2
malaise (General disorders) | 2
pyrexia (General disorders) | 5
hepatic function abnormal (Hepatobiliary disorders) | 2
seasonal allergy (Immune system disorders) | 2
gastroenteritis (Infections and infestations) | 6
hordeolum (Infections and infestations) | 5
impetigo (Infections and infestations) | 3
influenza (Infections and infestations) | 8
nasopharyngitis (Infections and infestations) | 14
oral herpes (Infections and infestations) | 3
pharyngitis (Infections and infestations) | 8
upper respiratory tract infection (Infections and infestations) | 14
contusion (Injury, poisoning and procedural complications) | 2
hand fracture (Injury, poisoning and procedural complications) | 2
joint sprain (Injury, poisoning and procedural complications) | 4
antinuclear antibody positive (Investigations) | 2
DNA antibody positive (Investigations) | 2
arthralgia (Musculoskeletal and connective tissue disorders) | 2
juvenile arthritis (Musculoskeletal and connective tissue disorders) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 2
headache (Nervous system disorders) | 3
cough (Respiratory, thoracic and mediastinal disorders) | 3
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
acne (Skin and subcutaneous tissue disorders) | 2
dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
dermatitis bullous (Skin and subcutaneous tissue disorders) | 2
eczema (Skin and subcutaneous tissue disorders) | 5
rash (Skin and subcutaneous tissue disorders) | 4
urticaria (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; the Medical Institution shall not disclose any material/information disclosed by Abbott Japan in connection with the Clinical Research or information obtained by conducting the Clinical Research to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting Clinical Research, Institution shall obtain Abbott Japan's prior written approval.